CLINICAL TRIAL: NCT02059642
Title: A 6-week Randomized, Multicenter, Double-blind, Parallel, Fixed-dose Study of MG01CI (Metadoxine Immediate-release/Slow-release, Bilayer Caplet) 1400 mg Compared With Placebo in Adults With Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: A 6 Week Study of MG01CI 1400 mg Compared With Placebo in Adults With ADHD ( Attention Deficit/Hyperactivity )
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alcobra Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL012
Record Dates: First submitted 2014-01-30; First posted 2014-02-11 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2014-03

CONDITIONS: ADHD; Attention-Deficit/Hyperactivity Disorder, Predominantly Inattentive Type
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet identical in appearance to study investigational product Route, frequency: Administered orally once daily
  Interventions: Drug: placebo
- MG01CI (1400 mg) (Experimental): MG01CI (Metadoxine Immediate-release/Slow-release, Bilayer Caplet) Dose, route, and frequency: 1400 mg administered orally once daily
  Interventions: Drug: MG01CI (1400 mg)

INTERVENTIONS:
Drug: MG01CI (1400 mg) — MG01CI (Metadoxine Immediate-release/Slow-release, Bilayer Caplet) 1400 mg administered orally once daily
  Other Names: Metadoxine Immediate-release/Slow-release, Bilayer Caplet
  Arms: MG01CI (1400 mg)
Drug: placebo — Placebo 1400 mg administered orally once daily
  Other Names: Inactive Drug
  Arms: Placebo

SUMMARY:
This study is a multisite, randomized, double-blind, placebo-controlled, phase 2/3 study of MG01CI (1400 mg daily) for 6 weeks compared with placebo in a 1:1 ratio of 300 adults with ADHD.

DETAILED DESCRIPTION:
This study is a multisite, randomized, double-blind, placebo-controlled, phase 2/3 study of MG01CI (1400 mg once daily) for 6 weeks compared with placebo in a 1:1 ratio of 300 adults with ADHD. The study comprises a Screening Visit at which initial assessment will be made and then a Washout Period during which prospective subjects must discontinue ADHD medication for 14 days (for psychotropic medications other than fluoxetine) or for 28 days (for fluoxetine) before randomization into the study. The Washout Period is 14 days, but may be extended to 28 days for a fluoxetine washout. Subjects requiring either a 14-day or a 28-day Washout Period will have an Interim Visit (off drug) on or about Day -8 (Day -10 to Day -3) for CAARS-Inv assessment after the Washout Period. The Baseline CAARS Inv assessment will be conducted on Day 0. If there is a ≥25% change in the CAARS-Inv results between the Interim Visit (off drug) assessment and the Baseline assessment, or if the subject does not return for the Baseline CAARS-Inv assessment, the subject will not be randomized. For subjects not needing washout, if there is a ≥25% change in the CAARS-Inv results between the Screening Visit assessment and the Baseline assessment, or if the subject does not return for the Baseline CAARS-Inv assessment, the subject will not be randomized. Following the Washout Period for those requiring a washout, or following the Screening Visit for those subjects who do not require a washout, eligible subjects will undergo baseline assessments and be randomized on Day 0 to MG01CI 1400 mg or to matching placebo and begin the Double-blind Treatment Period. The Double-blind Treatment Period will be 6 weeks in duration. There will be a 2-week Follow-up Period after the last dose of study treatment or early termination.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a man or a non-pregnant, non-lactating woman 18 to 55 years of age, inclusive, at the Screening Visit.
* Subject has a diagnosis of ADHD based on criteria in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) and DSM5.
* Subject has ADHD with at least moderate clinical severity (Clinical Global Impression-Severity [CGI-S]) score of 4 or greater).
* Subject has a score on the total ADHD symptom score with adult prompts of the CAARS-Inv of at least 22.
* Female subjects of childbearing potential must agree to use an effective contraceptive throughout the study
* Subject is able to attend the clinic regularly and reliably.
* Subject is able to swallow tablets and capsules.
* Subject is able to understand, read, write, and speak English fluently to complete the study-related materials (or Hebrew for Israeli subjects).
* Subject is able to understand and sign an informed consent form to participate in the study.

Exclusion Criteria:

* Subject did not respond in the past to 2 adequate trials of stimulant treatments or 1 adequate trial of atomoxetine treatment (in the investigator's judgment).
* Subject has any psychiatric condition clinically significant or unstable medical or surgical condition that may preclude safe and complete study participation as determined by the investigator .
* Subject has a known or suspected human immune deficiency virus-positive status or has diseases such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.
* Subject has a history of an allergy or sensitivity to B-complex vitamins.
* Subject has a history of intellectual disability or a history or suspicion of autism spectrum disorder.
* Subject has a current Axis I diagnosis (other than ADHD) according to the Structured Clinical Interview for DSM IV Axis I Disorders (SCID) or has a lifetime history of bipolar disorder or psychosis.
* Subject has used mega-dose vitamin B6/pyridoxine during the 28 days before the Screening Visit.
* Subject has used high-dose supplements of omega-3 fatty acids ≥ 500 mg on at least 1 day or folic acid supplements during the 2 weeks before the Screening Visit.
* Subject has used an investigational medication/treatment in the 30 days before the Screening Visit
* Subject has used any medication or food supplement that the investigator or the medical monitor considers unacceptable during the 14-day period before randomization.
* Subject has a current drug or alcohol dependence or substance abuse disorder according to DSM-IV. Subject should also agree to keep their caffeine intake consistent and refrain from consuming ≥300 mg per day of caffeine (no more than three 8-ounce servings of coffee) during the study.
* Subject has suicidality, defined as active ideation, an intent or plan, or any significant lifetime suicidal behavior. Subjects exhibiting history (within previous 12 months) of non-suicidal self-injurious behavior will be excluded.
* Subject has taken any prescription or non-prescription ADHD medications during the 14 days (for all psychotropic medications other than fluoxetine) or 28 days (for fluoxetine) before the randomization visit.
* Subject is significantly visually impaired to an extent that is not able to be corrected by prescription glasses or contact lenses
* Subject is related to the sponsor, investigator, or study staff.
* Subject has any condition that, in the principal investigator's opinion, would place the subject at risk or influence the conduct of the study or interpretation of results,
* Subject cannot fully comprehend the implications of the protocol, cannot comply with its requirements, or is incapable of following the study schedule for any reason.
* Subject is pregnant, lactating, or using an inadequate contraceptive method.
* If there is a ≥25% change in the CAARS-Inv results between the Interim visit (off drug) assessment and the Baseline assessment, or if the subject does not return for the Baseline CAARS-Inv assessment, the subject will not be randomized. For subjects not needing washout, if there is a ≥25% change in the CAARS-Inv results between the Screening Visit assessment and the Baseline assessment, or if the subject does not return for the Baseline CAARS-Inv assessment, the subject will not be randomized.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Weisler, MD, Principal Investigator — University of North Carolina, Duke University
Locations (20):
- United States (18):
  - Sarkis Clinical Trials, Gainesville, Florida
  - Miami Research, South Miami, Florida
  - Capstone Clinical Research, Libertyville, Illinois
  - Psychiatric Associates, Overland Park, Kansas
  - University Kentucky Psychiatry, Lexington, Kentucky
  - Pediatric Psychopharmacology & Adult ADHD Program, Massachusetts General Hospital, Boston, Massachusetts
  - Rochester Center For Behavioral Medicine, Rochester Hills, Michigan
  - Behavioral Medicine Center, Troy, Michigan
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - Bioscience Research, Mount Kisco, New York
  - Duke University, Durham, North Carolina
  - Richard H Weisler, MD, PA, Raleigh, North Carolina
  - Sequoia Behavioral Healthcare, Media, Pennsylvania
  - FutureResearch Trials, Austin, Texas
  - FutureResearch Trials Dallas, LP, Dallas, Texas
  - Bayou City Research, Houston, Texas
  - NeuroScience, Inc. (NSI), Herndon, Virginia
- Israel (2):
  - Neurocognitive unit Rambam MC, Haifa
  - ADHD unit Geha MC, Petah Tikva

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MG01CI (1400 mg)
Started | 148 | 152
Completed | 121 | 128
Not Completed | 27 | 24

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one dose of study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MG01CI (1400 mg) | Total
Number analyzed (Participants) | 146 | 152 | 298
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 146 | 152 | 298
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.42) | 35.1 (9.93) | 35.4 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 158
  Male | 67 | 73 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 10 | 25
  Not Hispanic or Latino | 131 | 141 | 272
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 130 | 128 | 258
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 105 | 108 | 213
  Israel | 41 | 44 | 85
BMI [Mean (Standard Deviation); unit: "kg/m^2"] | 28.243 (6.3923) | 28.345 (27.230) | 28.295 (6.3393)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total ADHD Symptom Score With Adult Prompts of the Conners Adult ADHD Rating Scale:O-SV in ADHD Adults From Baseline to 6 Weeks
Description: Primary efficacy endpoint: change from Baseline in the total ADHD symptom score with adult prompts of the CAARS-Inv. The CAARS is a scale to assess the presence and severity of ADHD symptoms and behaviors in adults. During an interview with the investigator, subject rates items pertaining to their behavior using a 4-point Likert-style format ranging from 0 ('Not at all') to 3 ('Very much). The scale measures ADHD symptoms across clinically significant domains using a 30 item questionnaire, while examining the manifestations of those symptoms. The scale includes an assessment of 9 inattentive symptoms (Subset A) and 9 hyperactive & impulsive symptoms (Subset B). The total ADHD symptom score, Subset C (the sum of the inattentive symptom scores from Subset A and the hyperactive & impulsive symptoms from Subset B) is the primary outcome measure. Scores of the scale for Subset C, comprised of scores from 18 questions,range from 0 (no ADHD symptoms) to 54, highest rating of ADHD symptoms.
Time Frame: baseline, 6 weeks
Population: Intent to Treat
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in Score from Baseline
Arm/Group | Placebo | MG01CI (1400 mg)
Number analyzed (Participants) | 146 | 151
Change in Score from Baseline | -9.9 [-11.89 to -7.92] | -12.0 [-13.95 to -10.06]
Statistical Analysis 1: Comparison: Placebo vs MG01CI (1400 mg); Test type: Superiority or Other; p = 0.1358, Mixed Models Analysis; MMRM: Model of Repeated Measures; Least Square Mean Difference = -2.10, 95% CI 2-sided [-4.87 to 0.66]

2. Secondary Outcome: Safety Evaluation of Treatment on the Basis of Percentage of Participants With Treatment Emergent Adverse Events
Description: Safety assessments will be based on changes from Baseline of clinical AEs reported by the subject or observed by the Investigator and concomitant medication use, treatment adherence (eg, dropouts due to AEs)
Time Frame: 6 weeks
Population: Safety population
Measure: Number; unit: Percentage of participants with TEAEs
Arm/Group | Placebo | MG01CI (1400 mg)
Number analyzed (Participants) | 146 | 152
Percentage of participants with TEAEs | 66.4 | 56.8

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Placebo | MG01CI (1400 mg)
Serious Adverse Events (participants affected / at risk) | 1/146 | 0/152
Other Adverse Events (participants affected / at risk) | 41/146 | 55/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=146) | MG01CI (1400 mg) (N=152)
APPENDICITIS (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=146) | MG01CI (1400 mg) (N=152)
NAUSEA (Gastrointestinal disorders) | 9 (9) | 13 (13)
FATIGUE (General disorders) | 12 (12) | 11 (11)
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 (2) | 8 (8)
HEADACHE (Nervous system disorders) | 18 (18) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"Publication of the Study results in scientific literature is encouraged, but any publication should require gaining prior approval from the Company and the Company reserves the right to review any paper written utilizing data generated from the Study before such paper is presented or submitted for publication".